CLINICAL TRIAL: NCT06576102
Title: Evaluation of Prevalence and Risk Factors of Persistent SARS-CoV-2 Infection in Immunocompromised Patients
Brief Title: Evaluation of Prevalence and Risk Factors of Persistent COVID-19 in Immunocompromised Patients
Acronym: PERsiCO
Status: Active, not recruiting | Type: Observational
Sponsor: Maddalena Giannella (Other)
Responsible Party: Sponsor-Investigator, Maddalena Giannella, Professor, University of Bologna
Organization: University of Bologna (Other)
Other Study IDs: PERsiCO
Record Dates: First submitted 2024-08-27; First posted 2024-08-28 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Persistent COVID-19; B Cell Malignancies
Keywords: COVID-19; Persistent SARS-CoV-2 infection; Immunocompromised patients; B cell malignancies; B cell targeting therapies; viral infections in the hematological patient
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with B cell malignancies: All immunocompromised adults (≥18 years) with a new SARS-CoV-2 infection assessed during the study period, hospitalized or followed as outpatients in the participating centers, will be screened for inclusion.
  Inclusion Criteria:
  * Diagnosis of B cell malignancies or previous treatment with B cell targeting therapies.
  * Diagnosis of proven SARS-CoV-2 infection confirmed by a PCR test (only the first infection during the study period will be considered, re-infection will be counted as a secondary endpoint).
  Interventions: Other: Persisting SARS-CoV-2 infection

INTERVENTIONS:
Other: Persisting SARS-CoV-2 infection — Prevalence of persisting SARS-CoV-2 infection among immunocompromised patients defined as the persistence or the recurrence of symptoms and signs (fever, dyspnea, hypoxemia, changes on chest-X ray or CT scan) and positive SARS-CoV-2 PCR ≥ 21 days after the time 0 (day of the first test positive for SARS-CoV-2 infection)

SUMMARY:
Spontaneous international multicenter retrospective and prospective observational study which objective is to evaluate the prevalence and risk factors of persistent SARS-CoV-2 infection within a population of hematology patients with humoral immunity deficiency.

DETAILED DESCRIPTION:
Spontaneous international multicenter retrospective and prospective observational study which objective is to evaluate the prevalence and risk factors of persistent SARS-CoV-2 infection within a population of hematology patients with humoral immunity deficiency.

The retrospective recruitment period will span from January, 1st, 2022 to the date of authorisation by hospital directorates following the Ethics Committees' approvals. This period has been established considering the prevalent diffusion of the omicron variant and its subvariants, which has led to significant changes in the clinical manifestations of COVID-19. The prospective recruitment will be carried out over the 12 months immediately following the retrospective period. During the study period, screening for persisting SARS-CoV-2 infection and therapeutic management of all patients will be carried out by the attending physicians according to routine practice.

This study is enclosed in the EU Horizon 2020 project "Connecting European Cohorts to Increase Common and Effective Response to SARS-CoV-2 Pandemic: ORCHESTRA" (Grant Agreement No. 101016167) and is located within Task 4.6 "Prevalence, risk factors and therapeutic management of persistent COVID-19 in frail patients." It is expected to enroll approximately 1,000 patients (500 at the coordinating center).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B cell malignancies or previous treatment with B cell targeting therapies.
* Diagnosis of proven SARS-CoV-2 infection confirmed by a PCR test (only the first infection during the study period will be considered, re-infection will be counted as a secondary endpoint).
* Provision of signed and dated informed consent.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All immunocompromised adults (≥18 years) with a new SARS-CoV-2 infection assessed during the study period, hospitalized or followed as outpatients in the participating centers, will be screened for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of persisting SARS-CoV-2 infection among immunocompromised patients | Retrospective recruitment period will span from January 1st, 2022 to to the date of authorisation by hospital directorates following the Ethics Committees' approvals
  The first primary endpoint variable will be the rate of patients with persisting SARS-CoV-2 infection among study patients with new diagnosis of SARS Cov2 during the study period Persisting COVID19 will be defined as the persistence or the recurrence of symptoms and signs (fever, dyspnea, hypoxemia, changes on chest-X ray or CT scan) and positive SARS-CoV-2 PCR ≥ 21 days after the time 0 (day of the first test positive for SARS-CoV-2 infection)

SECONDARY OUTCOMES:
Risk factors for persisting COVID19 | Retrospective recruitment period will span from January 1st, 2022 to to the date of authorisation by hospital directorates following the Ethics Committees' approvals
  Univariate and multivariate analysis will be carried out to investigate factors associated with persisting COVID-19 among the study population
Duration of viral shedding | Retrospective recruitment period will span from January 1st, 2022 to to the date of authorisation by hospital directorates following the Ethics Committees' approvals
  Duration of viral shedding, defined as the number of days between the first positive test and first negative PCR test
Duration of symptoms | Retrospective recruitment period will span from January 1st, 2022 to to the date of authorisation by hospital directorates following the Ethics Committees' approvals
  Duration of symptoms, defined as the number of days between symptoms onset and the clinical cure
Prevalence of imaging alterations | Retrospective recruitment period will span from January 1st, 2022 to to the date of authorisation by hospital directorates following the Ethics Committees' approvals
  Prevalence of imaging alterations, defined as the presence of new ground-glass and/or crazy paving and/or interstitial infiltrates at chest CT scan during the persisting infection (starting from 21 days after the first positive test until viral clearance)
Re-infection within 120 days | Retrospective recruitment period will span from January 1st, 2022 to to the date of authorisation by hospital directorates following the Ethics Committees' approvals
  Re-infection within 120 days, define as new positive test with or without symptoms after viral clearance has been achieved
All-cause 120-day mortality | Retrospective recruitment period will span from January 1st, 2022 to to the date of authorisation by hospital directorates following the Ethics Committees' approvals
  All-cause 120-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena Giannella, MD PhD, Principal Investigator — University of Bologna
Locations (5):
- Italy (4):
  - Irccs Aoubo, Bologna
  - IRCCS Humanitas, Milan
  - IRCCS INMI L. Spallanzani, Roma
  - AOUI Verona, Verona
- Hospital Virgen Macarena, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Since the study is conducted within the European Union's Horizon 2020 project named "ORCHESTRA" (grant agreement No 101016167), which will end on 30 November 2024, raw data will be available only after the end of the EU H2020 project on reasonable request

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT06576102/Prot_SAP_000.pdf